CLINICAL TRIAL: NCT04768192
Title: Functional and MRI Evaluation of the Robot-assisted and Traditional Rehabilitation Programs on the Muscle in Subjects With Acquired Brain Injury
Brief Title: Functional and MRI Evaluation of the Robot-assisted and Traditional Rehabilitation Programs on the Muscle
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS Eugenio Medea (Other)
Collaborators: The National Research Council, Italy (Other Government)
Responsible Party: Sponsor
Other Study IDs: GIP-745
Record Dates: First submitted 2021-02-18; First posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric patients with acquired brain injury: Subjects with a acquired brain injury occurred in the last 10 months prior the beginning of the treatment
  Interventions: Procedure: Physical Rehabilitation without lokomat; Procedure: Physical Rehabilitation with Lokomat

INTERVENTIONS:
Procedure: Physical Rehabilitation without lokomat — Conventional physiotherapy is performed in 10 weekly sessions (45 minutes each) over 4 weeks(total 40 sessions).
  Specific exercises are administered to improve gait, balance and functional abilities focusing on:
  strengthening the gluteus and quadriceps muscles stretching the hip flexor and hamstrings muscles increasing static balance increasing dynamic balance increasing functional abilities improving ground gait going up and down the stairs.
  Physiotherapists can choose from a list of 25 standard exercises, according to some constraints:
  1. strengthening exercises had to involve all the lower limb joints (no segmental intervention)
  2. during each session, at least 4 out of the 7 categories above had to be delivered
  3. the impossibility to perform any of the categories above during any session had to be recorded in the patient's treatment diary.
  Physiotherapists of the treatments group discuss patients' diaries during weekly meetings.
  Other Names: Conventional physiotherapy
Procedure: Physical Rehabilitation with Lokomat — The rehabilitation protocol consists of 20 sessions of robotic training alternated with 20 sessions of conventional physiotherapy (CP). Each treatment is performed in 5 weekly sessions (45 minutes each) over 4 weeks.
  Robotic training aimed to recovery/improve walking capacity from the initial Gross Motor Function Classification System (GMFCS) level. It is performed using the Lokomat® (Hocoma AG, Volketswil, Switzerland) gait orthosis. Initial set ups includes 50% body weight unload, gait velocity adjusted on the patient individual capability (1.5 km/h on average) and 100% guidance force. Both weight unload and guidance force are gradually reduced across sessions according to patient recovery of muscle strength and allowing patients to work harden and move more freely.
  Children engagement, active participation and motivation were reinforced through frequent encouragement by therapists and performance feedback implemented in the exercise video-games.
  Other Names: Lokomat

SUMMARY:
Walk recovery is one of the goals of rehabilitation programs in patients with acquired brain injury.

Recent experiences have shown the effectiveness of rehabilitation programs including traditional physiotherapy in combination with robotic gait training systems (Lokomat).

In this context, MRI can be used to assess the treatment effects on the muscular tissue, providing useful clinical indications for the optimization of the rehabilitation programs on the basis of the damage extension and the muscle characteristics.

DETAILED DESCRIPTION:
Acquired brain injuries can lead to permanent physical, cognitive and psycho-social deficits. One of the primary objectives of rehabilitation in these patients is to recover the ability to walk, which is usually feasible in most patients, even in those with severe brain injuries.

Recent experiences have shown that the use of rehabilitative programs that include traditional physiotherapy in combination with robotic walking training systems (robotic-aided gait training - RAGT, Lokomat) are effective in improving the performance of pediatric patients with acquired brain injuries. Thanks to the partial or total support of the patient's weight and the robotic guidance that facilitates a physiological gait pattern, these systems allow intensive and reproducible training which, by stimulating brain neuroplasticity, can increase the chances of recovery. Alterations of strength, coordination, balance associated with structural changes of muscular tissue (e.g. atrophy, fibrosis, adipose substitution) are frequent and may, on the other hand, compromise the effectiveness of rehabilitation treatments.

There are currently no literature data regarding local effects on muscle tissue of such treatments in the pediatric population; in particular, it has not yet been documented how the muscle responds to the robotic treatment and whether it is possible to identify local indices able to correlate with the degree of performance and improvement of each patient. Magnetic Resonance Imaging (MRI) can be a useful tool for in-vivo measurement of the effects of these treatments on muscle tissue and provide clinical indications for a better optimization of rehabilitative programs, based on the extent of damage and the characteristics of the muscle.

A complete evaluation of the effects of rehabilitative programs with RAGT, both in terms of mechanical-functional data (kinematics, muscular metabolism) and structural data through MRI, and the subsequent correlation of these parameters with clinical scales measuring motor skills, is not currently described in the literature. It could instead prove to be very useful both for prognostic purposes and for a better understanding of the local mechanisms of muscle tissue response to rehabilitative treatments, favoring an identification of the best rehabilitation plan targeted for each specific patient and thus increasing the chances of functional recovery.

The objectives of the study are:

1. To characterize, in subjects with acquired cerebral lesions, the effects of intensive rehabilitative programs with RAGT, in terms of kinematics, activation and muscle metabolism;
2. To document, in subjects with acquired cerebral lesions, the effects of intensive rehabilitative programs with RAGT on muscular structure through advanced and quantitative MRI methods;
3. Correlate functional and muscle imaging data with clinical parameters related to patient's motor skills and with the type of treatment performed.

ELIGIBILITY:
Inclusion Criteria:

* acquired brain lesion occurred in the last 10 months prior the beginning of the treatment
* hemi or tetraparesis diagnosis following the brain lesion
* thigh-bone length > 21 cm
* ability and willingness to follow instructions and communicate fear and pain

Exclusion Criteria:

* severe contractures, fractures, bone instability or osteoporosis of the lower limbs
* skin lesions in the lower limbs
* thromboembolic or cardiovascular pathologies
* aggression and self-aggressive behavior
* orthopedic surgery and/or botulinum toxin injection in the 6 months prior to enrollment
* cognitive and/or motor deficits prior to the injury
* contraindications to MRI examination

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population includes pediatric patients with acquired brain lesion occurred in the last 10 months prior the beginning of the treatment and showing deficit in the lower limbs movements due to the acquired lesion.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
GMFM - T-pre | The week before the beginning of the treatment
  Gross Motor Function Measures (GMFM) acquired before the beginning of the treatment. (Functional measure)
6mwt - T-pre | The week before the beginning of the treatment
  Six minute walking test (6mwt) performed before the beginning of the treatment. (Functional measure)
Ashowrth scale - T-pre | The week before the beginning of the treatment
  Ashowrth scale acquired before the beginning of the treatment. (Functional measure)
Tardieu scale - T-pre | The week before the beginning of the treatment
  Tardieu scale acquired before the beginning of the treatment. (Functional measure)
GMFM - T-post | Within a week after the ent of the treatment
  Gross Motor Function Measures (GMFM) acquired after the end of the treatment. (Functional measure)
6mwt - T-post | Within a week after the ent of the treatment
  Six minute walking test (6mwt) performed after the end of the treatment. (Functional measure)
Ashowrth scale - T-post | Within a week after the ent of the treatment
  Ashowrth scale acquired performed after the end of the treatment. (Functional measure)
Tardieu scale - T-post | Within a week after the ent of the treatment
  Tardieu scale acquired performed after the end of the treatment. (Functional measure)

SECONDARY OUTCOMES:
WF - T-pre | The week before the beginning of the treatment
  Water fraction (WF) in the muscular bundles measured from MRI Dixon data acquired before the beginning of the treatment
FF - T-pre | The week before the beginning of the treatment
  Fat fraction (FF) in the muscular bundles measured from MRI Dixon data acquired before the beginning of the treatment
FA - T-pre | The week before the beginning of the treatment
  Fractional Anisotropy (FA) in the muscular bundles measured from MRI Diffusion data acquired before the beginning of the treatment
MD - T-pre | The week before the beginning of the treatment
  Mean Diffusivity (MD) in the muscular bundles measured from MRI Diffusion data acquired before the beginning of the treatment
WF - T-post | Within a week after the end of the treatment
  Water fraction (WF) in the muscular bundles measured from MRI Dixon data acquired at the end of the treatment
FF - T-post | Within a week after the end of the treatment
  Fat fraction (FF) in the muscular bundles measured from MRI Dixon data acquired at the end of the treatment
FA - T-post | Within a week after the end of the treatment
  Fractional Anisotropy (FA) in the muscular bundles measured from MRI Diffusion data acquired at the end of the treatment
MD - T-post | Within a week after the end of the treatment
  Mean Diffusivity (MD) in the muscular bundles measured from MRI Diffusion data acquired at the end of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Denis Peruzzo, PhD, Principal Investigator — Research Institute IRCCS Eugenio Medea
Locations (1):
- Scientific Institute IRCCS Eugenio Medea, Bosisio Parini, LC, Italy

IPD SHARING:
Plan to Share IPD: No